CLINICAL TRIAL: NCT02074202
Title: A Phase III, Multi-center, Single-blind, Cross-over Study to Evaluate the Efficacy and Safety of 18Ffluorocholine (18F-FCH) Comparing With 18F-fluorodeoxyglucose (18F-FDG) for Detecting Hepatocellular Carcinoma
Brief Title: To Evaluate the Efficacy and Safety of (18F-FCH) Comparing With (18F-FDG) for Detecting Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201111019MIB
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Hepatocellular Carcinoma; Liver Disease
Keywords: 18F fluorocholine; 18F fluorodeoxyglucose; hepatocellular carcinoma; PET CT scan
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases | interventions — fluorocholine; Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCH PET/CT scan results (Experimental): PET/CT scan results with FCH intravenous injection
  Interventions: Drug: 18F- fluorocholine
- FDG PET/CT scan (Active Comparator): PET/CT scan results with FDG intravenous injection
  Interventions: Drug: 18F- fluorodeoxyglucose

INTERVENTIONS:
Drug: 18F- fluorocholine — To compare the diagnostic efficacy of FCH PET scan to FDG PET scan.
  Arms: FCH PET/CT scan results
Drug: 18F- fluorodeoxyglucose — To compare the diagnostic efficacy of FCH PET scan to FDG PET scan
  Arms: FDG PET/CT scan

SUMMARY:
Liver cancer is a major cause of death among patients of east or southeast asian descent, as well as other population groups, notably in central and west Africa. Diagnosis of liver cancer requires a combination of several imaging techniques and biopsies. Despite this, diagnosis can remain inconclusive or difficult to establish in patients at risk for liver cancer.

The purpose of this multi-center trial is to evaluate novel imaging methods developed to diagnose the most common form of liver cancer, hepatocellular carcinoma. We propose to use novel imaging probes that have been reported to bind to liver cancers but not benign liver lesions that can be confused with liver cancer. Two such imaging probes will be evaluated. 2-[18F]-fluoro-2-deoxy-D-glucose, called [18F]FDG, is a radioactive sugar that is widely used for cancer imaging with a device called positron emission tomography, or PET scans. We already know that [18F]FDG cannot detect some liver cancers that are slow growing. [18F]Fluorocholine ([18F]FCH), another molecule, has been recently reported to be highly effective at detecting liver cancer. In 2010, a French researcher reported 80-90% detection rate by using [18F]FCH alone or in combination with [18F]FDG.

We will compare [18F]FCH and [18F]FDG in evaluating 150 patients over a period of two years. The results will be correlated with those of biopsies and clinical follow-up.

This study will provide valuable data on whether these imaging agents can successfully differentiate malignant liver lesions from benign ones. It will also provide information about whether these imaging agents can successfully assess whether the cancer has spread outside the liver. It will provide data that will allow physicians to determine the optimal imaging protocol to properly diagnose liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 20 years old.
2. Patient who accepts to enter the study by signing written informed consent.
3. Patient with performance status ≤ 2 Eastern Cooperative Oncology Group (ECOG).
4. Patient with cirrhosis or chronic liver diseases suspected to have at least 1 hepatic nodule larger than 1 cm in diameter detected by conventional image (US, CT, MRI). Patient who has not yet received any therapy relevant to the aforementioned diagnosis. Hepatic nodule is defined as any one of the following conditions: suspicious hepatocellular carcinoma, benign tumor such as hemangioma, adenoma or focal nodular hyperplasia, metastatic lesions from other primary malignancy.
5. Female patient must take reliable contraception method(s) during the participation of the study.

Exclusion Criteria:

1. Patient has serious allergic history or known allergy to 18F-FDG or 18F-FCH.
2. Patient has been diagnosed of multiple malignancies.
3. Female patient who is pregnant, lactating or planning to become pregnant during the study.
4. Patient has been participated in other investigational trials within 28 days prior to study enrollment.
5. Patient is unable to undergo PET/CT scan.
6. Subjects with active systemic infections, or medical conditions that may significantly affect action, adequate uptake and elimination of radiotracer.
7. Subject with conditions judged by the investigator as unsuitable for the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The pathological diagnosis of the liver tumor will be compared with the test result of the PET/CT scan findings. | Within 6 months of follow up after the PET/CT scans.
  After the study cases finished the two PET/CT scans, the cases will be followed as long as 6 months thereafter. Within this time frame, the study cases will go for a patho-histological diagnosis of the liver tumor. This will be used as the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Yuan Tzen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan